CLINICAL TRIAL: NCT03935126
Title: A Biomarker Evaluation Study in Patients With Geographic Atrophy Secondary to Age-related Macular Degeneration (AMD) Evaluating the Use of Microperimetry (Fundus-controlled Perimetry) and Swept Source-OCT in Assessing Changes in Retinal Sensitivity and Anatomy Over Time.
Brief Title: Global Atrophie Biomarker Evaluation Study (GABiE)
Acronym: GABiE
Status: Terminated | Type: Observational
Why Stopped: Not due to safety reasons
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 0352-2110
Record Dates: First submitted 2019-04-30; First posted 2019-05-02 (Actual); Results first posted 2021-05-21 (Actual); Last update posted 2021-05-21 (Actual); Status verified 2021-04

CONDITIONS: Age-related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — Rapid Diagnostic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All patients
  Interventions: Diagnostic Test: Diagnostics

INTERVENTIONS:
Diagnostic Test: Diagnostics — Diagnostics

SUMMARY:
To investigate the use of microperimetry and SS-OCT in assessing the natural changes of retinal sensitivity and anatomy in the perilesional zone of geographic atrophy areas in patients with dry age-related macular degeneration.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated written informed consent in accordance with ICH-GCP and local legislation prior to admission to the study
* Age >=60 years
* Ability (including a sufficient general health status according to investigators judgement) and willingness to undertake all scheduled visits and assessments including predefined methodology and standards utilizing microperimetry GA secondary to AMD with no evidence of prior or active choroidal neovascularization (CNV) in the study eye
* GA lesion in the study eye must reside completely within the FAF imaging field (Field 2- 30 degree image centered on the fovea)
* BCVA of 20/63 or better (Snellen equivalent) using ETDRS charts at starting distance of 4 m in the study eye
* Well demarcated area(s) of GA secondary to AMD with no evidence of prior or active CNV in the study eye

  * The total GA lesion size >=1.2 mm^2 (approximately >=0.5 disc area [DA]) and <=17.78 mm^2 (approximately <=7 DA) and must reside completely within the FAF imaging field (Field 2-30 degree image centered on the fovea)
  * If GA is multifocal, at least 1 focal lesion must be >=1.2 mm^2 (approximately >=0.5 DA)
* Sufficiently clear ocular media, adequate pupillary dilation, and fixation to permit quality fundus imaging in the study eye

Exclusion Criteria:

* GA in either eye due to causes other than AMD (for example, monogenetic macular dystrophies [e.g., Stargardt disease, cone rod dystrophy] or toxic maculopathies [e.g., chloroquine/hydroxychloroquine maculopathy])
* Receiving active treatment in any studies of investigational drugs for GA/dry AMD in the study eye
* Mean sensitivity difference > 3 dB between the two microperimetry examinations in the screening visit.
* History of vitrectomy surgery, submacular surgery, or other surgical intervention for AMD in the study eye
* Previous laser photocoagulation for CNV, diabetic macular edema, retinal vein occlusion, and proliferative diabetic retinopathy in the study eye
* Prior treatment with Visudyne ®, external-beam radiation therapy, or transpupillary thermotherapy in the study eye
* History of prophylactic subthreshold laser treatment for AMD in the study eye
* Further criteria apply.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Geographic Atrophy (GA) secondary to Age-related Macular Degeneration (AMD) who are not receiving treatment for GA and have not previously receiving active treatment in clinical trials in the indication under invesitigation will be enrolled and followed for up to 12 months.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2019-05-07 (Actual); Primary Completion 2020-05-06 (Actual); Study Completion 2020-05-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Tufts Medical Center, Boston, Massachusetts, United States
- University Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder; 2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; 3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).
  For more details refer to: http://trials.boehringer-ingelheim.com/

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A biomarker evaluation study in patients with geographic atrophy secondary to age-related macular degeneration (AMD) evaluating the use of microperimetry (fundus-controlled perimetry) and Swept Source-Optical Coherence Tomography in assessing changes in retinal sensitivity and anatomy over observation period of 48 weeks.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria.
  Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- All Enrolled: All enrolled participants who had geographic atrophy secondary to age-related macular degeneration, signed informed consent for this trial, and met all inclusion criteria and none of the exclusion criteria, for evaluating the usage of microperimetry and Swept Source - Optical Coherence Tomography (SS-OCT) in assessing the natural changes of retinal sensitivity and anatomy in the retina. Each participant was planned to be observed for an observation period of 48 weeks after screening visit. During the observation period, 4 visits were planned to be taken at Week 0, 12, 24, and 48 of the observation period.
Period: Overall Study
Arm/Group | All Enrolled
Started | 3
Completed | 0
Not Completed | 3
Not completed — Study termination by sponsor | 3

BASELINE CHARACTERISTICS:
Population: Enrolled set: This subject set includes all subjects that signed informed consent for this trial.
Arm/Group | All Enrolled
Number analyzed (Participants) | 3
Age, Continuous [Mean (Standard Deviation); unit: Years] | 83.7 (4.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Retinal Sensitivity in the Junctional Zone and in the Perilesional Zone of the Largest Atrophic Loci as Assessed by Microperimetry for the Evaluation of Macular Functional Response at Week 12
Time Frame: At baseline and at week 12.
Population: Study was terminated early. 3 subjects were enrolled but no subject was entered. No outcome measures data was collected.
Arm/Group | All Enrolled
Number analyzed (Participants) | 0

2. Primary Outcome: Change From Baseline in Retinal Pigment Epithelium (RPE) Layer Thickness in the Junctional Zone and in the Perilesional Zone as Measured by Swept Source - Optical Coherence Tomography (SS-OCT) at Week 12
Time Frame: At baseline and at week 12.
Population: Study was terminated early. 3 subjects were enrolled but no subject was entered. No outcome measures data was collected.
Arm/Group | All Enrolled
Number analyzed (Participants) | 0

3. Primary Outcome: Change From Baseline in Photoreceptor Layer Thickness in the Junctional Zone and in the Perilesional Zone as Measured by Swept Source - Optical Coherence Tomography (SS-OCT) at Week 12
Time Frame: At baseline and at week 12.
Population: Study was terminated early. 3 subjects were enrolled but no subject was entered. No outcome measures data was collected.
Arm/Group | All Enrolled
Number analyzed (Participants) | 0

4. Secondary Outcome: Change From Baseline in Retinal Sensitivity in the Junctional Zone and in the Perilesional Zone of the Largest Atrophic Loci as Assessed by Microperimetry at Week 24 and 48
Time Frame: At baseline and at week 24 and 48.
Population: Study was terminated early. 3 subjects were enrolled but no subject was entered. No outcome measures data was collected.
Arm/Group | All Enrolled
Number analyzed (Participants) | 0

5. Secondary Outcome: Change From Baseline in Retinal Pigment Epithelium (RPE) Layer Thickness in the Junctional Zone and in the Perilesional Zone as Measured by Swept Source - Optical Coherence Tomography (SS-OCT) at Week 24 and 48
Time Frame: At baseline and at week 24 and 48.
Population: Study was terminated early. 3 subjects were enrolled but no subject was entered. No outcome measures data was collected.
Arm/Group | All Enrolled
Number analyzed (Participants) | 0

6. Secondary Outcome: Change From Baseline in Photoreceptor Layer Thickness in the Junctional Zone and in the Perilesional Zone as Measured by Swept Source - Optical Coherence Tomography (SS-OCT) at Week 24 and 48
Time Frame: At baseline and at week 24 and 48.
Population: Study was terminated early. 3 subjects were enrolled but no subject was entered. No outcome measures data was collected.
Arm/Group | All Enrolled
Number analyzed (Participants) | 0

7. Secondary Outcome: Change From Baseline in the GA Area as Measured by Fundus Autofluorescence (FAF) at Week 12, 24 and 48
Time Frame: At baseline and at week 12, 24 and 48
Population: Study was terminated early. 3 subjects were enrolled but no subject was entered. No outcome measures data was collected.
Arm/Group | All Enrolled
Number analyzed (Participants) | 0

8. Secondary Outcome: Change From Baseline in Best Corrected Visual Acuity (BCVA) Score as Assessed by Early Treatment Diabetic Retinopathy Scale (ETDRS) Chart at a Starting Distance of 4 Meters at Week 12, 24 and 48
Time Frame: At baseline and at week 12, 24 and 48.
Population: Study was terminated early. 3 subjects were enrolled but no subject was entered. No outcome measures data was collected.
Arm/Group | All Enrolled
Number analyzed (Participants) | 0

9. Secondary Outcome: Change From Baseline in Low Luminance Visual Acuity (LLVA) Score as Assessed by ETDRS Chart Under Low Luminance Conditions at a Starting Distance of 4 Meters at Week 12, 24 and 48
Time Frame: At baseline and at week 12, 24 and 48.
Population: Study was terminated early. 3 subjects were enrolled but no subject was entered. No outcome measures data was collected.
Arm/Group | All Enrolled
Number analyzed (Participants) | 0

10. Secondary Outcome: Number of Scotomatous Points Assessed by Microperimetry at Week 12, 24 and 48
Time Frame: At week 12, 24 and 48
Population: Study was terminated early. 3 subjects were enrolled but no subject was entered. No outcome measures data was collected.
Arm/Group | All Enrolled
Number analyzed (Participants) | 0

11. Secondary Outcome: Change From Baseline in the Area of Choroidal Non-perfusion as Measured Via Optical Coherence Tomography Angiography (OCT-A) at Week 12, 24 and 48
Time Frame: At baseline and at week 12, 24 and 48.
Population: Study was terminated early. 3 subjects were enrolled but no subject was entered. No outcome measures data was collected.
Arm/Group | All Enrolled
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From screening visit 1 until early termination of the study, up to 6 month + 5 days.
Description: Enrolled set: This subject set includes all subjects that signed informed consent for this trial.
Arm/Group | All Enrolled
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

LIMITATIONS AND CAVEATS:
Study was terminated early by the sponsor. No outcome measures data was collected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results.

Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days.

BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-21): https://cdn.clinicaltrials.gov/large-docs/26/NCT03935126/Prot_SAP_000.pdf